CLINICAL TRIAL: NCT04650984
Title: A Phase III Study Comparing the Efficacy of the Combination of Doxorubicin and the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF to Doxorubicin Alone as First-line Therapy in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: A Study Comparing the Efficacy of L19TNF+Doxorubicin vs Doxorubicin Alone as First-line Therapy in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Acronym: FIBROSARC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFDOX2-03/16
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Patients will receive 75 mg/m2 doxorubicin once every 3 weeks (reference treatment).
  Interventions: Drug: Doxorubicin
- Arm 2 (Experimental): Patients will receive 13 µg/kg L19TNF on days 1, 3 and 5 every 3 weeks in combination with 60 mg/m2 doxorubicin (once every 3 weeks).
  Interventions: Drug: Onfekafusp alfa; Drug: Doxorubicin

INTERVENTIONS:
Drug: Onfekafusp alfa — Patients will receive a fixed dose of L19TNF in combination with a fixed dose of doxorubicin.
  Other Names: L19TNF
  Arms: Arm 2
Drug: Doxorubicin — Patients will receive a fixed dose doxorubicin, administered as a 15 ± 5 minutes i.v. infusion.

SUMMARY:
The present study is an open-label, randomized, controlled, two-arm multi-center study of the efficacy of L19TNF treatment in combination with doxorubicin versus doxorubicin alone in advanced or metastatic soft-tissue sarcoma patients.

In the study, 102 patients will be randomized in a 1:1 ratio to receive doxorubicin treatment (Arm 1) or L19TNF treatment in combination with doxorubicin (Arm 2).

The primary objective of the trial is to evaluate if L19TNF in combination with doxorubicin (Arm 2) given for unresectable or metastatic soft tissue sarcoma improves efficacy measured as progression free survival, as compared to doxorubicin alone (Arm 1).

DETAILED DESCRIPTION:
Phase III, open label, randomized, controlled study in subjects with advanced or metastatic soft tissue sarcoma. In the study, 102 patients will be enrolled and parallel assigned in a 1:1 fashion to one of two different arms, as follows:

* ARM 1: Patients will receive 75 mg/m2 doxorubicin once every 3 weeks (reference treatment).
* ARM 2: Patients will receive 13 µg/kg L19TNF on days 1, 3 and 5 every 3 weeks in combination with 60 mg/m2 doxorubicin (once every 3 weeks).

Anti-cancer activity will be assessed every 6 weeks during therapy and every 12 weeks thereafter. Median PFS, PFS rates at 3, 6, 9, 12 and 18 months, mOS, OS rate at 12 and 18 months and ORR will be calculated.

Safety assessment will be performed on an ongoing basis during study participation, including standard laboratory assessments. The incidence of AEs will be summarized by severity in all patients with at least one study drug intake.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years.
2. Patients must have histological evidence of advanced unresectable and/or metastatic high-grade soft tissue sarcoma (grade 2 - 3 according to the FNCLCC grading system) not amenable to curative treatment with surgery or radiotherapy and for which doxorubicin treatment is considered appropriate. Participants with Osteosarcoma, Chondrosarcoma, Ewing Sarcoma/ Primitive Neuroectodermal Tumor (PNET), Kaposi's Sarcoma, Dermatofibrosarcoma protuberans, and Gastrointestinal Stromal Tumors (GIST) will be excluded
3. Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria 1.1. This lesion should not have been irradiated during previous treatments.
4. Life expectancy of at least 3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
6. Documented negative test for HIV-HBV-HCV. For HBV serology: the determination of HBsAg, anti-HBsAg-Ab and anti-HBCAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
7. Female patients: negative serum pregnancy test at screening for women of childbearing potential (WOCBP)*. WOCBP must agree to use, from the screening to six months following the last administration of L19TNF and/or Doxorubicin, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Male patients: Male subjects able to father children must agree to use two acceptable methods of contraception from the screening to four months following the last administration of L19TNF and/or Doxorubicin (e.g. condom with spermicidal gel). Double-barrier contraception is required.
8. Informed consent signed and dated to participate in the study.
9. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Prior therapy (except surgery and radiation) for unresectable or metastatic malignant soft tissue sarcoma.
2. Previous treatment with anthracycline-containing chemotherapy.
3. Radiotherapy within 4 weeks prior to therapy.
4. Known history of allergy to TNFα, anthracyclines or other intravenously administered human proteins/peptides/antibodies.
5. Previous therapy with recombinant TNF.
6. Absolute neutrophil count (ANC) < 1.5 x 109/L, platelets < 100 x 109/L and haemoglobin (Hb) < 9.0 g/dl.
7. Chronically impaired renal function or creatinine ≥ 2.0 x ULN.
8. Inadequate liver function (ALT, AST, ALP or total bilirubin ≥ 2.5 x ULN.
9. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
10. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
11. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
12. Clinically significant cardiac arrhythmias or requiring permanent medication.
13. Uncontrolled hypertension, despite optimal therapy.
14. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
15. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
16. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
17. Pregnancy or breast-feeding.
18. Requirement of chronic administration of corticosteroids or other immunosuppressant drugs. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
19. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
20. Known active or latent tuberculosis (TB).
21. Concurrent malignancies other than Soft Tissue Sarcoma, unless the patient has been disease-free for at least 2 years.
22. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
23. Serious, non-healing wound, ulcer or bone fracture.
24. Allergy to study medication or excipients in study medication.
25. Deep vein thrombosis, pulmonary embolism or other acute vascular events within 6 months.
26. Anticoagulation therapy with P2Y12 antagonists (e.g., clopidogrel, ticagrelor) and vitamin K antagonists (e.g., phenprocoumon, warfarin).
27. Concurrent use of other anti-cancer treatments or agents other than study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Median Progression free survival (mPFS) | From randomization up to week 72
  Progression-free survival PFS in a time-to-event analysis in the L19TNF plus Doxorubicin control group (Arm 2) versus the Doxorubicin alone treatment group (Arm 1).

SECONDARY OUTCOMES:
PFS rate | At 3, 6, 9, 12, 18 months after randomization
  Progression Free Survival
Overall Response Rate (ORR) | At 3, 6, 9, 12, 18 months after randomization
  Rate of Complete Response and Partial Response of L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1).
Overall survival (OS) | At 12 months and 18 months after randomization
  OS in the L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1)
Median Overall survival (mOS) | At 12 months and 18 months after randomization
  mOS in the L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1).
Adverse Events | From week 1 up to week 72
  Number of patients with adverse events (AEs) assessed on CTCAE v.4.03
HAFA assessment | At day 1 of week 1 and week 2; at day 1 from week 4 up to week 18, every 3 weeks; at week 22-23 (EoT); at week 23-24 (first follow-up visit)
  Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19TNF (Arm 2).

CONTACTS AND LOCATIONS:
Locations (28):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Charité- Universitätsmedizin Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinik Hamburg-Eppendorf, Hamburg
  - Heidelberg University Hospital, Heidelberg
  - Universitätsmedizin der J.-G. Universität Mainz, Mainz
  - Klinik rechts der Isar, München
  - Universitaetsklinikum Muenster, Münster
- Italy (4):
  - IRCCS Fondazione del Piemonte per l'Oncologia Istituto per la Ricerca e la Cura del Cancro di Candiolo, Candiolo, Torino
  - Bologna University, Chemotherapy Unit, IRCCS Istituto Ortopedico Rizzoli, Department of DIMES, Bologna
  - AOU San Luigi Gonzaga, Orbassano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Poland (2):
  - Szpital Pomorski Im. PCK, Gdynia
  - Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie Warszawa, Warsaw
- Spain (6):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Fundación Jiménez Díaz, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Miguel Servet, Zaragoza